CLINICAL TRIAL: NCT00826995
Title: Comparison of Video-based Versus Written Patient Education on Melanoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 200816692-1
Record Dates: First submitted 2009-01-20; First posted 2009-01-22 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Melanoma; Malignant Melanoma
Keywords: patient Education; dermatology Patient Education; melanoma; melanoma education; malignant melanoma; melanoma detection
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Video-based education arm: (Experimental): Subjects receiving the video-based educational material
  Interventions: Other: Patient Educational Materials
- Written education arm: (Active Comparator): Subjects receiving the written educational material
  Interventions: Other: Patient Educational Materials

INTERVENTIONS:
Other: Patient Educational Materials — In the experimental arm, the intervention is the video-based patient educational material on melanoma. In the active comparison arm (control arm), the comparison intervention is written patient educational material on melanoma.
  Other Names: Patient educational materials on melanoma detection

SUMMARY:
The purpose of this study is to compare the effect of video-based patient education with written instruction on subjects' understanding of melanoma.

DETAILED DESCRIPTION:
We plan to conduct a randomized, controlled trial comparing the effect of video-based patient education with written instruction on subjects' understanding of melanoma.

Subjects randomized to the video-based education arm will be instructed to watch a video on the definition of melanoma, risk factors associated with the development of melanoma, and signs that should prompt an evaluation for melanoma. Subjects randomized to the written education arm will receive written information on the definition of melanoma, risk factors associated with the development of melanoma, and signs that should prompt an evaluation for melanoma. The contents of the video and the written educational materials will be comparable.

At the end of the study period 1 month later, subjects will be interviewed via telephone regarding their understanding of melanoma. Subjects will also be interviewed regarding their comprehension and attitude towards video-based and written education materials.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older at time of consent, may be men or women.
* Able to adhere to the study visit schedule and other protocol requirements.
* Capable of giving informed consent.

Exclusion Criteria:

* Non-English speaking individuals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2009-01; Primary Completion 2009-05 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Knowledge of melanoma detection. | 1 month

SECONDARY OUTCOMES:
Subjects' comprehension and attitude towards video-based and written education materials. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: April W Armstrong, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Department of Dermatology, Sacramento, California, United States

REFERENCES:
- See also: University of California-Davis Department of Dermatology Clinical Research — http://www.ucdmc.ucdavis.edu/dermatology/research/clinical